CLINICAL TRIAL: NCT03976037
Title: Buccal Versus Vaginal Misoprostol In Combination With Foley Bulb for Labor Induction at Term: a Randomized Controlled Trial
Brief Title: Buccal Versus Vaginal Misoprostol In Combination With Foley Bulb
Acronym: BEGIN
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Christiana Care Health Services (Other)
Responsible Party: Principal Investigator, Helen Beatriz Gomez, Resident Physician, Christiana Care Health Services
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DDD# 604291
Record Dates: First submitted 2019-05-31; First posted 2019-06-05 (Actual); Last update posted 2021-02-26 (Actual); Status verified 2021-02

CONDITIONS: Induction of Labor
MeSH Terms: interventions — Misoprostol

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vaginal Misoprostol in combination with foley bulb (Active Comparator): Women in the vaginal misoprostol-cervical Foley group will have both misoprostol and a cervical Foley placed. Patients will receive 25 micrograms of misoprostol per vagina along with the insertion of a16F Foley catheter with a stylet. The Foley balloon catheter will be filled with 30cc balloon inserted digitally or by direct visualization with a speculum. The Foley bulb will be placed just above the level of the internal os and inflated with 30cc of sterile water.
  Vaginal misoprostol can be repeated up to five additional times for a maximum of 24 hours or a total of 6 doses if the patient is not contracting more than 3 times per 10 minutes. If the patient is contracting more than 3 times per 10 minutes after 6 hours, oxytocin protocol is initiated.
  Interventions: Drug: Misoprostol
- Buccal Misoprostol in combination with foley bulb (Active Comparator): misoprostol and a cervical Foley placed. Patients will receive 25 micrograms of buccal misoprostol along with the insertion of a16F Foley catheter with stylet. The Foley balloon catheter will be filled with 30cc balloon inserted digitally or by direct visualization with a speculum. The Foley bulb will be placed just above the level of the internal os and inflated with 30cc of sterile water.
  Buccal misoprostol can be repeated up to five additional times for a maximum of 24 hours or a total of 6 doses if the patient is not contracting more than 3 times per 10 minutes. If the patient is contracting more than 3 times per 10 minutes after 6 hours, oxytocin protocol is initiated.
  Interventions: Drug: Misoprostol

INTERVENTIONS:
Drug: Misoprostol — Women randomized to either vaginal or buccal misoprostol-cervical Foley group will have both misoprostol and a cervical Foley placed. Patients will receive 25 micrograms of vaginal or buccal misoprostol along with the insertion of a16F Foley catheter with stylet. The Foley balloon catheter will be filled with 30cc balloon inserted digitally or by direct visualization with a speculum. The Foley bulb will be placed just above the level of the internal os and inflated with 30cc of sterile water.
  vaginal or Buccal misoprostol can be repeated up to five additional times for a maximum of 24 hours or a total of 6 doses if the patient is not contracting more than 3 times per 10 minutes. If the patient is contracting more than 3 times per 10 minutes after 6 hours, oxytocin protocol is initiated.
  Other Names: cytotec

SUMMARY:
Combined misoprostol and Foley bulb catheter has been shown to be an effective induction method. However, optimal route of administration for misoprostol has not been established.

Therefore, the purpose of this study is to compare the effectiveness and safety of combination buccal miso-foley to combination vaginal miso-foley for third trimester cervical ripening and induction of labor.

DETAILED DESCRIPTION:
This randomized controlled trial of consenting women undergoing induction of labor with combined misoprostol and Foley catheter seeks to efficacy of vaginal versus buccal misoprostol route of administration.

This project will include 216 women presenting at Christiana Care Health System. Women will be included if they are at least 37 weeks gestation, have a singleton pregnancy, have intact membranes and are undergoing an induction of labor using a Foley catheter combined with misoprostol. Following admission, women will be randomized into either vaginal or buccal misoprostol.

Women will be randomized with equal probability to the intervention group using block randomization stratified by party.

Patients will receive 25 micrograms of misoprostol along with the insertion of a16F Foley catheter. Misoprostol can be repeated up to five additional times for a maximum of 24 hours or a total of 6 doses if the patient is not contracting more than 3 times per 10 minutes. The remainder of labor management will be at the discretion of each woman's obstetric provider.

Prior to discharge from the hospital, baseline demographic and clinical data will be obtained via chart review

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* full term (≥37 weeks) gestations determined by routine obstetrical guidelines
* singleton gestation in cephalic presentation
* Both nulliparous and multiparous women
* Intact membranes
* Cervical dilation ≤2cm

Exclusion Criteria:

* Any contraindication to a vaginal delivery or to misoprostol
* fetal demise
* Multifetal gestation
* prior uterine surgery, previous cesarean section
* Tachysystole was defined as at least 6 contractions in 10 minutes for 2 consecutive 10-minute periods
* women with HIV, and women with medical conditions requiring an assisted second stage
* Additional exclusion criteria were as follows: category 3 fetal heart rate tracing, hemolysis elevated liver enzymes and low platelets (HELLP) syndrome or eclampsia, growth restriction <10th percentile (based on Hadlock growth curves) with reversal of flow in umbilical artery Doppler studies, and growth restriction <5th percentile with elevated, absent, or reversal of flow in umbilical artery Doppler studies

As described in previous research (Levine LD, Downes KL, Elovitz MA, Parry S, Sammel MD, Srinivas SK. Mechanical and Pharmacologic Methods of Labor Induction: A Randomized Controlled Trial. Obstet Gynecol. 2016;128(6):1357-1364)

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 216 (Actual)
Dates: Start 2019-06-04 (Actual); Primary Completion 2020-01-20 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
time to delivery (hours) defined | through study completion, an average of 2 year
  as time from initiation of induction method to delivery time, regardless of mode of delivery.

SECONDARY OUTCOMES:
Rate of Cesarean delivery | through study completion, an average of 2 year
  yes/no
Time to active labor | through study completion, an average of 2 year
  s time from initiation of induction method to dilatation ≥6cm
Maternal length of stay | through study completion, an average of 2 year
  defined as length of time from admission for induction to discharge postpartum, days
Indication for cesarean delivery | through study completion, an average of 2 year
  The reason for induction: NRFHT, arrest of dilation, arrest of descent, failed IOL, other
Rate of 3rd/4th degree perineal laceration | through study completion, an average of 2 year
  yes/no
Rate of Maternal Blood transfusion | through study completion, an average of 2 year
  yes/no
Rate of Endometritis | through study completion, an average of 2 year
  yes/no; fundal tenderness and fever that required treatment with antibiotics
Rate of Wound separation-infection | From time of delivery to time of hospital discharge; up to 6 weeks
  the need for additional wound closure or the need for antibiotics
Rate of Venous thromboembolism | through study completion, an average of 2 year
  yes/no
Rate of Hysterectomy | through study completion, an average of 2 year
  yes/no
Rate of Intensive care unit admission | through study completion, an average of 2 year
  yes/no
Rate of Maternal Death | through study completion, an average of 2 year
  yes/no
Rate of Chorioamnionitis | through study completion, an average of 2 year
  the presence of maternal fever ≥100·4°f in the presence of maternal or fetal tachycardia or fundal tenderness
Rate of terbutaline use | through study completion, an average of 2 year
  yes/no
Rate of Intrauterine pressure catheter use | through study completion, an average of 2 year
  yes/no
Rate of Amnioinfusion | through study completion, an average of 2 year
  yes/no
Rate of Analgesia use | through study completion, an average of 2 year
  yes/no
Rate of Severe respiratory distress syndrome | From time of delivery to hospital discharge; up to 6 weeks
  defined as intubation and mechanical ventilation for a minimum of 12 hours
Rate of Culture proven-presumed neonatal sepsis | From time of delivery to hospital discharge; up to 6 weeks
  yes/no
Rate of Neonatal blood transfusion | From time of delivery to hospital discharge; up to 6 weeks
  yes/no
Rate of Hypoxic ischemic encephalopathy | From time of delivery to hospital discharge; up to 6 weeks
  yes/no
Rate of Intraventricular hemorrhage grade 3 or 4 | From time of delivery to hospital discharge; up to 6 weeks
  yes/no
Rate of Necrotizing enterocolitis | From time of delivery to hospital discharge; up to 6 weeks
  yes/no
Rate of head cooling. | From time of delivery to hospital discharge; up to 6 weeks
  yes/no
Rate of NICU admission | From time of delivery to hospital discharge; up to 6 weeks
  yes/no

CONTACTS AND LOCATIONS:
Overall Officials: Helen B Gomez, MD, Principal Investigator — Christiana Care Health Services
Locations (1):
- Christiana Care Health Systems, Newark, Delaware, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Levine LD, Downes KL, Elovitz MA, Parry S, Sammel MD, Srinivas SK. Mechanical and Pharmacologic Methods of Labor Induction: A Randomized Controlled Trial. Obstet Gynecol. 2016 Dec;128(6):1357-1364. doi: 10.1097/AOG.0000000000001778. PMID 27824758
- [Background] Chung JH, Huang WH, Rumney PJ, Garite TJ, Nageotte MP. A prospective randomized controlled trial that compared misoprostol, Foley catheter, and combination misoprostol-Foley catheter for labor induction. Am J Obstet Gynecol. 2003 Oct;189(4):1031-5. doi: 10.1067/s0002-9378(03)00842-1. PMID 14586350
- [Derived] Gomez HB, Hoffman MK, Caplan R, Ruhstaller K, Young MHH, Sciscione AC. Buccal vs vaginal misoprostol combined with Foley catheter for cervical ripening at term (the BEGIN trial): a randomized controlled trial. Am J Obstet Gynecol. 2021 May;224(5):524.e1-524.e8. doi: 10.1016/j.ajog.2021.02.016. Epub 2021 Feb 19. PMID 33617796